CLINICAL TRIAL: NCT03716206
Title: Effects of Exergames on Post-stroke Shoulder Pain and Motor Function
Brief Title: Exergames on Shoulder Pain and Motor Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201810003B
Record Dates: First submitted 2018-10-20; First posted 2018-10-23 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Shoulder Pain; Stroke
Keywords: Shoulder Pain; Stroke; Motor function
MeSH Terms: conditions — Shoulder Pain; Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exergames group (Experimental): The exergames intervention is one hour per day, four or five days per week for three weeks.
  Interventions: Device: Exergame
- conventional group (Active Comparator): The conventional group intervention is one hour per day, four or five days per week for three weeks.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Device: Exergame — This intervention included upper limb task-orientation training, upper limb coordination training, shoulder range of motion and upper limb activity training.
  Arms: exergames group
Other: Physical therapy — This intervention included upper limb task-orientation training, upper limb coordination training, shoulder range of motion and upper limb activity training.
  Arms: conventional group

SUMMARY:
This study is to investigate the effects of exergame on shoulder pain and motor function of upper extremity in individuals with stroke.

DETAILED DESCRIPTION:
Background and Purpose: Stroke is a major cerebrovascular disorder causing various symptoms in the world. A substantial portion of those surviving from stroke typically experience neurological sequelae and stroke-related complications. Post stroke shoulder pain is a sensory disturbance is one of a common complication in patients with chronic stroke and may adversely affect patients' quality of life. Nowadays, exergame has been explored as an adjunct therapy for the management of pain for a number of conditions. This study is to investigate the effects of exergame on shoulder pain and motor function of upper extremity in individuals with stroke. Method: This is a randomized controlled trail. Sixty subjects with poststroke shoulder pain will be recruited and randomized into either the exergame (experimental) group or conventional (control) group. The intervention is one hour per day, four or five days per week for three weeks. The primary outcomes are Visual Analogue Scale, and Brief Pain Inventory - Short Form. The secondary outcomes are Fugl-Meyer Assessment for Upper Limb Extremity, Wolf motor function test and Shoulder Pain and Disability Index.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral hemiplegia caused by stroke
2. Modified Ashworth Scale ≤2。
3. Mini-Mental State Examination ≥24。
4. Age ≥20。
5. Shoulder pain 。

Exclusion Criteria:

1. Shoulder joint contructure
2. Forzen shoulder
3. Dizzness, lesion of auditory and vision.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - Short Form | Change from Baseline at 7 weeks
  To assess the severity of pain and the impact of pain on daily functions. The Brief Pain Inventory - Short Form assess severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week. It is available in a short (nine items) form.
Visual analogue scale | Change from Baseline at 7 weeks
  The VAS provides a continuous scale for magnitude estimation and consists of a straight line, the ends of which are defined in terms of the extreme limits of pain experience. VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (worst) to the right (best).

SECONDARY OUTCOMES:
Wolf motor function test | Change from Baseline at 7 weeks
  This test was designed to assess the motor ability of patients with moderate to severe upper extremity motor deficits in the laboratory and clinic. The WMFT tests a broad range of upper extremity function through two strength measurements and a series of 15 functional tasks that progress from simple movements in proximal joint areas to complex movements in distal joint areas. The final time score will be the median time required for all timed tasks executed. One hundred twenty seconds is the maximum time allowed for each task attempted.
Fugl-Meyer Assessment | Change from Baseline at 7 weeks
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. However, reflex activity is measured using 2 points only, with a score of 0 or 2 for absence and presence of reflex respectively. it is common practice to assess all domains separately. The Maximum score in upper limb is 66.

OTHER OUTCOMES:
Shoulder Pain Disability Index | Change from Baseline at 7 weeks
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou, Taiwan